CLINICAL TRIAL: NCT06844500
Title: Phase 3, Randomised Maternal and Infant (From 4 to 24 Months of Age) Safety and Immunogenicity Trial of MVA-BN® Vaccine in the Democratic Republic of the Congo
Brief Title: Phase 3 Maternal Safety & Immunogenicity Trial of MVA-BN® in DRC
Acronym: PregInPoxVac
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jean-Pierre Van geertruyden (Other)
Collaborators: PENTA Foundation (Network); Ace Africa (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Bavarian Nordic (Industry); University of Kinshasa (Other)
Responsible Party: Sponsor-Investigator, Jean-Pierre Van geertruyden, Prof. Dr, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PIPVac-001 Maternal component
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Neonate; Maternal Transmission; Mpox; Vaccination; Immunogenicity; Safety; Pregnancy; Postpartum
Keywords: MVA-BN vaccine; mpox; Monkeypox virus; Pregnant women; Newborn; Phase 3; Vaccine; Adults; Randomised; Open-label; Immune transfer; Paediatrics; Obstetrics; Gynaecology; Smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic; Neonate; adolescents
MeSH Terms: conditions — Mpox, Monkeypox; Smallpox

STUDY DESIGN:
Intervention Model Description: 359 healthy pregnant participants will be randomised (3:2) to receive the standard MVA-BN vaccine of two doses, administered 28 days apart, during pregnancy (N= 215), or in the immediate postpartum (N=144 ).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Maternal Group 1 (Active Comparator): Women in Maternal Group 1 (vaccination during pregnancy), will receive the first of two MVA-BN vaccine doses, subcutaneously, in the second or third trimester of pregnancy, yet before 32 weeks of gestation. Ideally, both doses are administered during pregnancy.
  Interventions: Biological: MVA-BN standard regimen
- Maternal Group 2 (Active Comparator): Women in Maternal Group 2 (vaccinated postpartum), will receive the first of two MVA-BN vaccine doses, subcutaneously, ≤72 hours after delivery, preferably before discharge from the hospital/maternal health clinic (if applicable), unless contraindicated by the gynaecologist.
  Interventions: Biological: MVA-BN standard regimen
- Maternal Group 3 (Active Comparator): Women exposed to clinically or laboratory-confirmed mpox cases (Maternal Group 3) will preferably be vaccinated within 4 days after exposure. However the vaccine will be provided until 14 days after exposure if no symptoms are present.
  Interventions: Biological: MVA-BN standard regimen (Administered as PEP)
- Historical Arm (Other): Historical data from healthy adults aged 18 to 50 years old from the POX-MVA-045 study (NCT06549530), will be used for safety and immunogenicity (non-inferiority) comparisons.
  Interventions: Biological: MVA-BN standard regimen

INTERVENTIONS:
Biological: MVA-BN standard regimen — The MVA-BN vaccine, with the active ingredient: Modified Vaccinia Ankara-Bavarian Nordic, will be administered as a standard two-dose regimen at 1x10^8 TCID50 Inf.U./0.5 mL. The doses will be given 28 days apart (±3 days) via subcutaneous injection into the deltoid muscle, preferably in the non-dominant arm.
  Arms: Historical Arm; Maternal Group 1; Maternal Group 2
Biological: MVA-BN standard regimen (Administered as PEP) — MVA-BN. Post Exposure Prophylaxis (PEP)
  The MVA-BN vaccine, with the active ingredient: Modified Vaccinia Ankara-Bavarian Nordic, will be administered as a standard two-dose regimen at 1x10^8 TCID50 Inf.U./0.5 mL. The doses will be given 28 days apart (±3 days) via subcutaneous injection into the deltoid muscle, preferably in the non-dominant arm.
  For Maternal Group 3, MVA-Bn will be administered as PEP as soon as possible after exposure, preferably within 4 days after exposure. However, as per WHO guidelines, PEP will be offered up to 14 days after exposure if the pregnant woman has not yet developed symptoms.
  Arms: Maternal Group 3

SUMMARY:
This Phase 3 open-label study aims to assess the safety and immune response of the MVA-BN mpox vaccine when administered subcutaneously to pregnant and postpartum women in the Democratic Republic of the Congo (DRC), a population at high risk of mpox infection. The study will be conducted in Boende, Tshuapa Province, DRC.

A total of 359 maternal participants, aged 16 to 35 and in their second or third trimester of pregnancy, will be enrolled. Participants will be randomly assigned to receive two subcutaneous doses of the MVA-BN vaccine, given 28 days apart, either during pregnancy (Maternal Group 1) or within 72 hours after delivery (Maternal Group 2). Additionally, pregnant women in any trimester who have been recently exposed to a confirmed mpox case will be enrolled in the post-exposure prophylaxis (PEP) arm (Maternal Group 3), receiving the vaccine as soon as possible after exposure-ideally within four days but up to 14 days if they remain asymptomatic.

The study will evaluate the safety, reactogenicity, and immune responses of vaccinated pregnant women compared to healthy adults in the POX-MVA-045 study (NCT06549530) through non-inferiority analyses. Participants will be monitored for immunogenicity and safety for 13 months post-delivery, while neonates will be observed for safety over the same period. The trial will also compare outcomes between women vaccinated during pregnancy and those vaccinated postpartum, assess the transfer of maternal immunity to neonates, and explore correlations between maternal antibody levels in serum and breast milk.

This study seeks to provide strong evidence supporting the safety and immunogenicity of the MVA-BN mpox vaccine in pregnancy, contributing to global public health efforts to protect at-risk women and their infants in mpox-endemic regions.

DETAILED DESCRIPTION:
This open-label, Phase 3 study aims to evaluate the immunogenicity and safety of the MVA-BN standard regimen (1x10⁸ TCID50 Inf.U./0.5mL) administered subcutaneously in two doses, 28 days apart, to pregnant women and women in the immediate postpartum period (<72 hours after delivery). As described in the study protocol, the main study consists of the vaccination and safety and immunogenicity follow-up of pregnant and postpartum women. A sub-study will evaluate the transmission of antibodies from mother to child either during pregnancy of via breast milk.

The trial plans to enrol 359 participants, aged 16 to 35 years, with a gestational age between 13 and 32 weeks. Participants will be randomised into three groups: Maternal Group 1 (N=215), vaccinated during pregnancy; Maternal Group 2 (N=144), vaccinated within 72 hours postpartum; and Maternal Group 3 (N=convenience sampling), which includes pregnant women exposed to a confirmed mpox case within the past 14 days but who remain asymptomatic and will be offered post-exposure prophylaxis (PEP).

The study will be conducted at the General Reference Hospital of Boende, located in Boende, Tshuapa Province, Democratic Republic of Congo (DRC), with two satellite sites (Motema Mosantu and Marie-Louise Health Centres) supporting maternal delivery, vaccination for Maternal Group 2, and immediate postpartum sample collection, where applicable.

During the screening visit (SCR), interested participants will undergo an evaluation (test of understanding) to ensure understanding of the study and provide informed consent (or assent for minors). Demographics, vaccination history, and medical history will be recorded. Participants' general health will be evaluated through a physical examination, urine testing, and a gynaecological ultrasound to confirm gestational age. Blood samples will be collected for haematology, biochemistry, and infection screening for HIV, hepatitis B, syphilis, and malaria. After enrolling participants will be randomised to Maternal Group 1 or Maternal Group 2, unless they have been exposed to mpox in the past 14 days, then they will enrolled in Maternal group 3. All AEs, including serious adverse events (SAEs), medically attended adverse events (MAAEs), and adverse events of special interest (AESIs), will be monitored from enrolment until 13 months after delivery.

The prenatal visits (PN) are scheduled according to gestational age: PN Visit 1 (15-18 weeks), PN Visit 2 (24-28 weeks), PN Visit 3 (28-32 weeks), and PN Visit 4 (36-38 weeks). The number of visits will depend on the participant's enrolment date. Where feasible and applicable, prenatal visits will be combined with screening and/or vaccination visits. At each visit, vital signs and anthropometric measurements (weight, height, and fundal height) will be recorded to monitor maternal health and foetal growth. Urinary tests for infections will be performed at each visit, and a glucose challenge test (GCT) at 24-28 weeks will screen for gestational diabetes. Ultrasounds will also be performed as needed to evaluate gestational health. All participants will receive Intermittent Preventive Treatment for malaria (IPTp) according to WHO guidelines, with doses spaced at least one month apart.

On Day 0, participants' vital signs (blood pressure, heart rate, respiratory rate, and temperature) will be assessed. Blood samples will be collected from mothers to establish baseline immunogenicity, including neutralising antibodies (PRNTs), total binding antibodies (ELISA), and IgG binding antibodies (LUMINEX assay) against vaccinia and mpox viruses. To minimise inconvenience and where possible and applicable, samples for haematology and biochemistry will be collected simultaneously. Afterwards, participants will receive their first dose of the MVA-BN vaccine and a participant journal to record any solicited or unsolicited adverse events (AEs).

Seven days after the first vaccine dose (Day 0), the participant will be asked to return with the journal to record data on solicited AEs and unsolicited AEs (UAEs). Ongoing solicited AEs at this visit will be followed up until resolution and UAEs will be followed up until 28 days post-vaccination and inquired about before the second vaccine dose.

On Day 28, physical examinations of the mother will be conducted. Participants will receive the second MVA-BN vaccine dose, and blood samples will be collected from mothers to measure neutralising antibodies (PRNTs), total binding antibodies (ELISA), and IgG binding antibodies (LUMINEX assay). Participants will also receive a second participant journal to record any AEs.

Seven days after the first vaccine dose (Day 35), the participant will be asked to return with the journal to record data on solicited AEs and unsolicited AEs (UAEs). Ongoing solicited AEs at this visit will be followed up until resolution and UAEs will be followed up until 28 days post-vaccination during a telephone or home visit on Day 56.

On Day 42, blood samples will be collected from mothers to evaluate the persistence of vaccine-induced antibodies.

On Day 56, ongoing solicited AEs will be followed up and any ongoing or new UAEs be assessed/followed up via telephone or home visit.

On delivery day (Dd), a cord blood sample will be collected to measure neutralising antibodies (PRNTs), total binding antibodies (ELISA), and IgG binding antibodies (LUMINEX assay). Within 72 hours postpartum, colostrum (breast milk) samples will be collected to measure IgA antibody levels using the LUMINEX assay, reflecting maternal immunity transfer through breastfeeding. Physical examinations of both the mother and neonate will be conducted. Neonatal assessments will include APGAR scores at 1 and 5 minutes, general appearance, measurements (weight, length, and head circumference), and reflexes. Maternal assessments will focus on recovery and any postpartum complications. Maternal Group 2 will be vaccinated within 72 hours postpartum with the first MVA-BN dose, this will be Day 0 for this Group. All other visits from Day 0-Day 56 will take place for this group as described above. The Day 42 visit corresponds with the 6 week post-partum visit. Activities for both visits will be combined in to one visit.

Post-delivery visits will occur at 6 weeks, 12 weeks, 6 months and 13 months post delivery for all participants. Mothers and neonates will undergo follow-up assessments, including physical examinations of neonates to evaluate growth and developmental milestones. Blood samples will be collected from mothers at each visit to monitor the durability of vaccine-induced antibodies. Additionally, breast milk samples will be collected on at 6 weeks, 12 weeks, 6 months and 13 months post delivery to evaluate IgA binding antibody levels. At 6 weeks and 12 weeks postpartum visits, IgG binding antibodies in breast milk will also be determined. Blood samples from neonates will be collected on at 6 weeks, 12 weeks and 6 months after birth to assess neutralising antibodies (PRNTs), total binding antibodies (ELISA), and IgG binding antibodies (LUMINEX assay).

ELIGIBILITY:
Inclusion Criteria:

1. The participant must be between 16 and 35 years of age inclusive on the consent day.
2. The participant must pass (≥9/10) the Test of Understanding after being advised of the risks and benefits of the trial in a language understood by the participant and before performing any trial-specific procedures.

   * Note: For participants 16-17 years old, the parent/legal guardian must also pass the test of understanding.
   * Note: If the participant or parent/legal guardian for 16-17-year-olds fails the TOU test on the first attempt, he/she must be retrained on the purpose of the study and must take the test again (2 repeats are allowed). If participants or their parent/legal guardian fail on the third attempt, they should not continue with screening or consenting procedures.
   * Note: Maternal Group 3 participants are not restricted to 3 attempts to pass the TOU. For ethical reasons, these participants will be offered unlimited attempts.
3. The participant must sign and date an informed consent form (≥18 years old) or assent form (16-17 years old) indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study.

   * Note: If the participant is under 18 years of age, informed consent must also be obtained from a parent/legal guardian capable of providing consent. The consent form must be signed and dated by the parent/guardian after they have read and understood the risks and benefits of the trial and before any trial-specific procedures are performed.
   * Note: The partner (father of the child) or guardian for the follow-up of the infant after delivery) must also sign an informed consent/assent form (ICF) indicating that they understand the purpose of, and procedures required for, the study and is willing for their child to participate in the study.
   * Note: In case the participant, partner, parent/legal guardian cannot read or write, the procedures must be explained in the presence of an impartial (i.e. not involved in the study) third party witness, and informed consent must be obtained from this impartial third party witness.
4. The participant must be in her second (13-27 weeks) or early third trimester (28-32 weeks) of pregnancy at the time of vaccination.

   - Note: Mpox-infected and exposed pregnant women (Maternal group 3) can enrol at any stage of the pregnancy.

   - Note: Depending on enrolment progress of pregnant women between 13 and 32 weeks gestation, pregnant women in their first trimester may be enrolled but will not be vaccinated until they reach 13 weeks gestation. Sponsor approval needs to be sought to start enrolling pregnant women earlier than 13 weeks gestation.
5. The participant and her unborn child must be generally healthy in the investigator's clinical judgment and on the basis of vital signs assessed at day 1 screening with no severe (chronic) conditions (as far as medically known) that might interfere with vaccine assessment.

   - Note: HIV-positive subjects can be enrolled as long as their general condition is good, i.e., HIV infection under stable Highly Active Antiretroviral Therapy (HAART; no change within the last three month) and/or CD4 count >500/ μL, no signs or symptoms of immunosuppression. Pregnant HIV-positive participants must agree to attend all prenatal visits foreseen in the time and events schedule for regular follow-up.
   * Note: HBV-positive pregnant women will receive treatment according to the National guidelines and can be enrolled as long as their general condition is good. The decision to enrol falls under the discretion of the PI.
   * Note: Participants who test positive for syphilis at screening can be reassessed for enrolment after treatment has been provided.
6. The participant must be pregnant with a singleton pregnancy.
7. The participant must live in the Boende health zone or its surrounding health zones in the Tshuapa province of the DRC.
8. The participant must be willing to deliver her child to the General Referral Hospital of Boende (the trial site location) or the satellite sites Motema Mosantu Health Centre or Marie-Louse Health Centre or the participant must be willing to inform the study staff when labour has started (either through the GRH or satellite site staff, through family or via mobile phone).
9. The participant must agree to follow the study protocol, including attending follow-up visits and reporting delivery plans and any adverse events.
10. The participant must be available and willing to participate and for her unborn child to participate for the duration of the study.
11. The participant must be willing to provide verifiable identification, such as iris scanning or a participant card where feasible, and have means to be contacted (phone number or address).

Inclusion criteria for the Maternal Group 3:

1. Close contact in the 2 weeks prior to signing the ICF with anyone known to have mpox.

Exclusion Criteria:

1. Known history of cowpox, mpox or vaccinia infection.
2. Close contact in the 2 weeks before signing the ICF with anyone known to have mpox.

   - Note: not applicable to Maternal Group 3
3. Known history of or active autoimmune disease (vitiligo or thyroid disease requiring thyroid replacement are not exclusions), history of Guillain-Barré syndrome or Reye's syndrome.
4. Having received any smallpox or licensed or investigational poxvirus-based (e.g. ACAM2000, MVA-BN based like MVA-BN-Filo) vaccine in the past.
5. Must not have received another experimental or non-licensed vaccine within 4 weeks before receiving the MVA-BN vaccine and during the trial.
6. Known allergy or history of anaphylaxis or other severe adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines), including known allergy to egg, egg products and aminoglycosides.
7. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g., tris(hydroxymethyl)-amino methane, including a history of allergic asthma.
8. Acute or chronic medical condition that, in the opinion of the investigator, would render the trial procedures unsafe or would interfere with the evaluation of responses, including but not limited to neurologic, cardiovascular, respiratory, hepatic, hematologic, rheumatologic, endocrine, gastrointestinal, renal, autoimmune, or immunosuppressive conditions.

   - Note: Participants with minor acute illnesses such as mild diarrhoea or mild upper respiratory tract infection or temperature ≥38.0ºC at screening will be excluded from enrolment at that time but may be rescheduled for re-screening later if feasible.
9. Presence of significant medical conditions or clinically significant findings at screening or vital signs for which, in the opinion of the gynaecologist/medical doctor, participation would not be in the best interest of the participant (e.g., compromise the safety or well-being) or that could prevent, limit, or confound the protocol-specified assessments.

   * Note: Participants who have recently received treatment for acute, uncomplicated malaria are eligible for participation if at least 3 days have elapsed from the conclusion of a standard, recommended course of therapy for malaria; participants who are acutely ill with malaria at the time of screening should complete therapy and wait an additional 3 days after completion before screening for the study.
   * Note: Participants with sickle cell trait can be included.
10. History of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision at least 6 months prior to screening that is considered to have achieved cure
11. Clinically significant mental disorder not adequately controlled by medical treatment.
12. Active or recent (within 6 months before screening) chronic alcohol abuse and/or intravenous and/or nasal drug abuse.
13. Recent blood donation (including platelets, plasma, and red blood cells) within 4 weeks before screening or planned blood donations during the active trial period.
14. Chronic systemic administration (defined as more than 14 days) of >5 mg prednisone (or equivalent)/day or any other immune-modifying drugs from 3 months before the first trial vaccination to the visit at the end of the active trial period (use of topical, inhaled, ophthalmic, and nasal glucocorticoids is allowed).

    - Note: Participants receiving antiretroviral (ARV) medication for the management of HIV infection are eligible for inclusion, provided they meet inclusion criterion 5.
15. History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, significant arrhythmia with or without corrective/ablative surgery, or any other heart condition under the care of a doctor.
16. Major surgery (per the investigator's judgment) within the 4 weeks before screening or planned major surgery during the study (from the start of screening onwards).
17. Post-organ and/or stem cell transplant, whether or not with chronic immunosuppressive therapy.
18. Administration or planned administration of immunoglobulins and/or any blood products from 3 months prior to the first trial vaccination until the visit at the end of the active trial period (packed red blood cells given for an emergency indication in an otherwise healthy person and not required as ongoing treatment is not exclusionary [e.g., packed red blood cells given in an emergency during elective surgery])
19. Received an investigational or nonregistered drug or vaccine or used an invasive investigational or nonregistered medical device within 30 days prior to vaccination or current or planned participation in another clinical study during the study.

    - Note: Participation in an observational clinical study is allowed.
20. History of chronic urticaria (recurrent hives).
21. Employment with the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, or relationship to the investigator or study site employee.

Additional inclusion criteria for Maternal Group 3:

1. No symptoms at the time of reporting/vaccination.

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 359 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Main study: Neutralising antibody response post-dose 2 vaccination with MVA-BN | 14 days after the second dose
  To assess the immunogenicity of the MVA-BN standard regimen, administered SC, in eliciting neutralising antibodies against the vaccinia virus in women vaccinated during pregnancy compared to adults of the POX-MVA-045 study at 2 weeks after the second dose.
Safety and reactogenicity of the MVA-BN vaccine in pregnant women | Throughout the trial period; from first vaccination to 13 months postpartum.
  To assess the safety and reactogenicity of the MVA-BN standard regimen, administered SC, in pregnant women compared to adults of the POX-MVA-045 study.
Neonatal/infant safety outcomes in offspring of vaccinated mothers | Throughout the trial period; from delivery to 13 months postpartum.
  To assess the safety in neonates/infants born to mothers vaccinated during pregnancy and mothers vaccinated postpartum.
Maternal, fetal, and neonatal outcomes in vaccinated women | From vaccination to 13 months postpartum
  To describe maternal, foetal and neonatal outcomes in the cohort vaccinated during pregnancy, compared to the cohort vaccinated postpartum (control) and, if possible, the outcomes of pregnancy surveillance in Boende for the duration of the study.
Sub-study. Maternal immunity transferred via breastmilk | At delivery
  To assess immunogenicity in infants at birth by measuring the amount of total binding antibodies against the vaccinia virus, neutralising antibodies against the vaccinia virus, IgG binding antibodies against the vaccinia and mpox viruses in cord blood from women vaccinated during pregnancy compared to women vaccinated in the postpartum.
Immunogenicity in maternal serum post-vaccination | Baseline to 13 months postpartum
  To assess the immunogenicity in mothers of the MVA-BN standard regimen, administered SC, in eliciting IgG binding antibodies against vaccinia and monkeypox virus in maternal blood from women vaccinated during pregnancy compared to women vaccinated in the postpartum at baseline (prior to vaccination), 2 weeks after the second dose, at delivery (when not the same as baseline), and at 6 weeks, 12 weeks, 6 months, and 13 months postpartum.
Maternal immunity transferred via breastmilk (IgA antibodies) | Delivery to 13 months postpartum
  To assess maternal immunity transferred via breastmilk by measuring IgA binding antibodies against vaccinia and monkeypox virus in breastmilk samples from women vaccinated during pregnancy compared to women vaccinated in the postpartum period in colostrum, at 6 weeks, 12 weeks, 6 months and 13 months postpartum.
Maternal immunity transferred via breastmilk (IgG antibodies) | 6 weeks and 12 weeks postpartum
  To assess maternal immunity transferred via breastmilk by measuring IgG binding antibodies against vaccinia and monkeypox virus in breastmilk samples from women vaccinated during pregnancy compared to women vaccinated in the postpartum period at 6 weeks and 12 weeks postpartum.
Persistence of maternal immunity in infants | 6 weeks to 6 months postpartum
  To assess persistence of maternal immunity in infants by measuring neutralising antibodies against the vaccinia virus, total binding antibodies against the vaccinia virus, IgG binding antibodies against vaccinia and monkeypox viruses in the infant's blood born from women vaccinated during pregnancy compared to women vaccinated in the postpartum at 6 weeks, 12 weeks, and 6 months postpartum.

SECONDARY OUTCOMES:
Neutralising antibody response in women vaccinated during pregnancy and adult of the POX-MVA-045 study | Baseline to 13 months postpartum
  To assess the immunogenicity of the MVA-BN standard regimen, administered SC, in eliciting neutralising antibodies against the vaccinia virus in women vaccinated during pregnancy compared to adults of the POX-MVA-045 study at baseline and all blood collection time points after the second dose.
Neutralising antibody response in women vaccinated in the immediate postpartum and adult of the POX-MVA-045 study | Delivery to 13 months postpartum
  To assess the immunogenicity of the MVA-BN standard regimen, administered SC, in eliciting neutralising antibodies against the vaccinia virus in women vaccinated in the immediate postpartum period compared to adults of the POX-MVA-045 study at baseline and all blood collection time points after the second dose.
Neutralising antibody response in women vaccinated during pregnancy and women vaccinated in the immediate postpartum | Baseline to 13 months postpartum
  To assess the immunogenicity of the MVA-BN standard regimen, administered SC, in eliciting neutralising antibodies against the vaccinia virus in women vaccinated during pregnancy compared to women vaccinated in the postpartum, at baseline, 6 weeks, 12 weeks, 6 months and 13 months after delivery.
Binding antibody reponse in women vaccinated during pregnancy and adults of the POX-MVA-045 study | Baseline to 13 months postpartum
  To assess the immunogenicity of the MVA-BN standard regimen, administered SC, in eliciting total binding antibodies against the vaccinia virus in women vaccinated during pregnancy compared to adults of the POX-MVA-045 study at baseline and all blood collection time points after the second dose.
Binding antibody reponse in women vaccinated in the immediate postpartum period and adults of the POX-MVA-045 study | Throughout the trial period; from first vaccination to 13 months postpartum
  To assess the immunogenicity of the MVA-BN standard regimen, administered SC, in eliciting total binding antibodies against the vaccinia virus in women vaccinated in the immediate postpartum period compared to adults of the POX-MVA-045 study at baseline and all blood collection time points after the second dose.
Binding antibody reponse in women vaccinated during pregnancy and women vaccinated in the immediate postpartum | Delivery to 13 months postpartum
  To assess the immunogenicity of the MVA-BN standard regimen, administered SC, in eliciting total binding antibodies against the vaccinia virus in women vaccinated during pregnancy compared to women vaccinated in the immediate postpartum period, at baseline, 2 weeks after the second dose, delivery, 6 weeks (if different from 2 weeks after the second dose), 12 weeks, 6 months and 13 months after delivery.
Safety and reactogenicity of the MVA-BN in women vaccinated in the immediate postpartum and adults of the POX-MVA-045 study | Throughout the trial period; from first vaccination to 13 months postpartum.
  To assess the safety and reactogenicity of the MVA-BN standard regimen administered to women in the immediate postpartum compared to adults (POX-MVA-045).
Safety and reactogenicity of the MVA-BN in women vaccinated during pregnancy and women vaccinated in the immediate postpartum | Throughout the trial period; from enrolment to 1 year after second dose
  To assess the safety and reactogenicity of the MVA-BN standard regimen administered in pregnant women compared to women in the immediate postpartum period.
Correlation between maternal IgG in serum and IgA antibody levels in breastmilk | From delivery to 13 months postpartum
  To explore whether there is a correlation between maternal IgG antibody levels against the vaccinia and mpox virus in serum and maternal IgA antibody levels against the vaccinia and mpox virus in breastmilk of women vaccinated during pregnancy or women vaccinated in the postpartum at delivery and at 6 weeks, 12 weeks, and 6 months, 13 months postpartum.
Correlation between maternal IgG antibody levels in serum and breastmilk in the first 12 weeks postpartum | 6 weeks and 12 weeks postpartum
  To explore whether there is a correlation between maternal IgG antibody levels against the vaccinia and mpox virus in serum and breastmilk of women vaccinated during pregnancy or women vaccinated in the postpartum at 6 and 12 weeks postpartum.
Correlation between maternal IgA and IgG antibody levels in breastmilk | Baseline to 13 months postpartum
  To explore whether there is a correlation of maternal IgA and IgG antibodies against the vaccinia and mpox virus in breastmilk in women vaccinated during pregnancy or women vaccinated in the postpartum at 6 weeks and 12 weeks.

OTHER OUTCOMES:
Immunogenicity of MVA-BN used as PEP in women exposed during pregnancy | Baseline to 13 months postpartum
  To assess the immunogenicity of the MVA-BN standard regimen, administered SC, in eliciting neutralising antibodies against the vaccinia virus in PEP women vaccinated during pregnancy compared to women not exposed to mpox and vaccinated during pregnancy at baseline, 2 weeks after the second dose, and at 6 weeks, 12 weeks, 6 months and 13 months after delivery.
Binding antibody response in PEP women vaccinated during pregnancy versus non-exposed women | Delivery to 13 months postpartum
  To assess the immunogenicity of the MVA-BN standard regimen, administered SC, in eliciting total binding antibodies against the vaccinia virus in PEP women vaccinated during pregnancy compared to women not exposed to mpox and vaccinated during pregnancy at baseline, 2 weeks after the second dose, and at and at 6 weeks, 12 weeks, 6 months and 13 months after delivery.
safety and reactogenicity of the MVA-BN in PEP women vaccinated during pregnancy | Throughout the trial period; from first vaccination to 13 months postpartum.
  To assess the safety and reactogenicity of the MVA-BN standard regimen, administered SC in PEP women vaccinated during pregnancy compared to women not exposed to mpox and vaccinated during pregnancy.
Safety in newborns/infants born to mothers vaccinated with PEP | From delivery to 13 months postpartum
  To assess safety in newborns/infants born to mothers vaccinated with PEP compared to those born to mothers vaccinated during pregnancy not exposed to mpox.
Pregnancy, foetal and neonatal outcomes | Baseline to 13 months postpartum
  To describe pregnancy and foetal, and neonatal outcomes in children born to PEP women compared to women not exposed to mpox and vaccinated during pregnancy (control) and, if possible, the outcomes of pregnancy surveillance in Boende for the duration of the study.
Demographic and obstetric variables impacting infant antibodies | From enrolment to 13 months postpartum
  To explore which demographic and obstetric variables (e.g. age, sex, gestational age at vaccination during pregnancy, malaria exposure, HIV status, malnutrition, etc.) impact the neutralising, total binding antibody, and IgG binding (as applicable) antibody response against the vaccine antigen in the serum of (exposed) pregnant and postpartum women and their newborn/infant.
Neutralising antibody response in a subset of women vaccinated during pregnancy and during the immediate postpartum | Baseline to 13 months postpartum
  To assess the immunogenicity of the MVA-BN standard regimen, administered SC, in eliciting neutralising antibodies against the monkeypox and vaccinia virus in a subset (10%) of women vaccinated during pregnancy compared to a subset (10%) of women vaccinated in the immediate postpartum period at baseline, 2 weeks after the second dose, at delivery, and 6 weeks (if different from 2 weeks after the second dose), 12 weeks, 6 months and 13 months after delivery.
Total IgG Response Against Multiple MPXV Antigens with Standard and Half-Dose Regimens. | Baseline to 13 months postpartum
  To assess the immunogenicity of the MVA-BN standard regimen, administered SC, in eliciting Total IgG in serum with multiple MPXV specific antigens (B6R, B2R, E8L, M1R, A35, H3L) in a subset (10%) of women vaccinated during pregnancy compared to a subset (10%) of women vaccinated in the immediate postpartum period at baseline, 2 weeks after the second dose, at delivery, and 6 weeks (if different from 2 weeks after the second dose), 12 weeks, 6 months and 13 months after delivery.
Demographic and obstetric variables impacting cord blood antibodies | Cord blood collected at delivery
  To explore which demographic and obstetric variables (e.g. age, sex, gestational age at vaccination during pregnancy, malaria exposure, HIV-status, malnutrition, etc.) impact the presence of maternally derived neutralising, total binding, and IgG binding antibodies against the vaccine antigen in cord blood.
Demographic and obstetric variables impacting breastmilk antibodies | Baseline to 13 months postpartum
  To explore which demographic and obstetric variables (e.g. age, sex, gestational age at vaccination during pregnancy, malaria exposure, malnutrition, etc.) impact the presence of maternally derived neutralising, total binding, and IgG and IgA binding antibodies against the vaccine antigen in breastmilk.
Impact of demographic variables on presence of maternally derived antibodies in infant's blood sample | Baseline to 13 months postpartum
  To explore which demographic and obstetric variables (e.g. age, sex, gestational age at vaccination during pregnancy, malaria exposure, malnutrition, etc.) impact the presence of maternally derived neutralising, total binding, and IgG and IgA binding antibodies against the vaccine antigen in infant's blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre Van geertruyden Van geertruyden, Prof. Dr, Study Director — Universiteit Antwerpen
Locations (1):
- Boende Hôpital Général de Référence, Boende, Province de La Tshuapa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lemey G, Lariviere Y, Zola TM, Maketa V, Matangila J, Mitashi P, Vermeiren P, Thys S, De Bie J, Muhindo HM, Ravinetto R, Van Damme P, Van Geertruyden JP. Algorithm for the support of non-related (serious) adverse events in an Ebola vaccine trial in the Democratic Republic of the Congo. BMJ Glob Health. 2021 Jun;6(6):e005726. doi: 10.1136/bmjgh-2021-005726. PMID 34183329
- [Background] Zola Matuvanga T, Lariviere Y, Lemey G, De Bie J, Milolo S, Meta R, Esanga E, Vermeiren PP, Thys S, Van Geertruyden JP, Van Damme P, Maketa V, Matangila J, Mitashi P, Muhindo-Mavoko H. Setting-up an Ebola vaccine trial in a remote area of the Democratic Republic of the Congo: Challenges, mitigations, and lessons learned. Vaccine. 2022 May 31;40(25):3470-3480. doi: 10.1016/j.vaccine.2022.04.094. Epub 2022 May 9. PMID 35550847
- [Background] Puri A, Pollard AJ, Schmidt-Mutter C, Laine F, PrayGod G, Kibuuka H, Barry H, Nicolas JF, Lelievre JD, Sirima SB, Kamala B, Manno D, Watson-Jones D, Gaddah A, Keshinro B, Luhn K, Robinson C, Douoguih M; EBL4001 Study Group. Long-Term Clinical Safety of the Ad26.ZEBOV and MVA-BN-Filo Ebola Vaccines: A Prospective, Multi-Country, Observational Study. Vaccines (Basel). 2024 Feb 17;12(2):210. doi: 10.3390/vaccines12020210. PMID 38400193
- [Background] Salloum M, Paviotti A, Bastiaens H, Van Geertruyden JP. The inclusion of pregnant women in vaccine clinical trials: An overview of late-stage clinical trials' records between 2018 and 2023. Vaccine. 2023 Nov 22;41(48):7076-7083. doi: 10.1016/j.vaccine.2023.10.057. Epub 2023 Oct 28. PMID 37903681
- [Background] Lariviere Y, Zola T, Stoppie E, Maketa V, Matangila J, Mitashi P, De Bie J, Muhindo-Mavoko H, Van Geertruyden JP, Van Damme P. Open-label, randomised, clinical trial to evaluate the immunogenicity and safety of a prophylactic vaccination of healthcare providers by administration of a heterologous vaccine regimen against Ebola in the Democratic Republic of the Congo: the study protocol. BMJ Open. 2021 Sep 28;11(9):e046835. doi: 10.1136/bmjopen-2020-046835. PMID 34588237
- [Background] Schwartz DA, Pittman PR. Mpox (Monkeypox) in Pregnancy: Viral Clade Differences and Their Associations with Varying Obstetrical and Fetal Outcomes. Viruses. 2023 Jul 28;15(8):1649. doi: 10.3390/v15081649. PMID 37631992
- [Background] Schwartz DA. High Rates of Miscarriage and Stillbirth among Pregnant Women with Clade I Mpox (Monkeypox) Are Confirmed during 2023-2024 DR Congo Outbreak in South Kivu Province. Viruses. 2024 Jul 13;16(7):1123. doi: 10.3390/v16071123. PMID 39066285
- [Background] Kozlov M. Monkeypox virus: dangerous strain gains ability to spread through sex, new data suggest. Nature. 2024 May;629(8010):13-14. doi: 10.1038/d41586-024-01167-5. No abstract available. PMID 38653833
- [Background] Bunge EM, Hoet B, Chen L, Lienert F, Weidenthaler H, Baer LR, Steffen R. The changing epidemiology of human monkeypox-A potential threat? A systematic review. PLoS Negl Trop Dis. 2022 Feb 11;16(2):e0010141. doi: 10.1371/journal.pntd.0010141. eCollection 2022 Feb. PMID 35148313
- See also: MVA-BN — https://www.bavarian-nordic.com/pipeline/technology/mva-bn.aspx
- See also: MVA-BN Product Characteristics — https://ec.europa.eu/health/documents/community-register/2022/20220722156674/anx_156674_en.pdf